CLINICAL TRIAL: NCT01917630
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study of the Efficacy and Safety of ALV003 Treatment in Symptomatic Celiac Disease Patients Maintained on a Gluten-Free Diet
Brief Title: Evaluation of the Efficacy and Safety of ALV003 in Symptomatic in Celiac Disease Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alvine Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALV003-1221
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Gluten-free diet; Coeliac disease; Celiac sprue
MeSH Terms: conditions — Celiac Disease | interventions — ALV003

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALV003 (Experimental)
  Interventions: Drug: ALV003
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ALV003 — ALV003 is an orally administered mixture of two enzymes (cysteine endoprotease B-isoform 2 and prolyl endopeptidase)
  Arms: ALV003
Drug: placebo
  Arms: Placebo

SUMMARY:
To determine the effects of 12 weeks administration of different dose levels of ALV003 on the mucosal lining of the small intestine and symptoms in celiac disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 80 years
* Physician diagnosed celiac disease
* Adherence to a gluten-free diet
* Experiencing symptoms of celiac disease over a 1-month period
* Willing to take study medication for 12 weeks
* Willing to comply with all study procedures
* Sign informed consent

Exclusion Criteria:

* Active inflammatory bowel disease
* Active dermatitis herpetiformis
* Use of certain specific medications prior to entry
* History of alcohol or illicit drug abuse in previous 6 months
* Pregnant or lactating
* Received any experimental drug within 30 days of enrollment
* Uncontrolled chronic disease or condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Intestinal mucosal morphometry | 12 weeks
  Change in villus height to crypt depth (Vh:Cd) ratio between baseline and week 12

SECONDARY OUTCOMES:
Efficacy: Intestinal intraepithelial lymphocyte density | 12 weeks
  Change in intestinal intraepithelial lymphocytes between baseline and week 12 (CD3+ cells/100 epithelial cells)
Safety: safety and tolerability of ALV003 | 12 weeks
  Incidence of adverse events between baseline and week 12

OTHER OUTCOMES:
Celiac disease-specific serology | 12 weeks
Quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Adelman, MD, Study Director — Alvine Pharmaceuticals Inc.
Locations (82):
- United States (73):
  - Decatur, Alabama
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Los Angeles, California
  - Modesto, California
  - Newport Beach, California
  - Oceanside, California
  - Orange, California
  - Palo Alto, California
  - Poway, California
  - Roseville, California
  - San Diego, California
  - San Jose, California
  - San Marcos, California
  - Aurora, Colorado
  - Bridgeport, Connecticut
  - Boynton Beach, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Largo, Florida
  - Miami, Florida
  - Naples, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Oak Lawn, Illinois
  - Des Moines, Iowa
  - Topeka, Kansas
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Boston, Massachusetts
  - Chesterfield, Michigan
  - Wyoming, Michigan
  - Rochester, Minnesota
  - Jackson, Mississippi
  - Kansas City, Missouri
  - Mexico, Missouri
  - Marlton, New Jersey
  - Great Neck, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Mentor, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Malvern, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Chattanooga, Tennessee
  - Hermitage, Tennessee
  - Houston, Texas
  - Irving, Texas
  - Southlake, Texas
  - West Jordan, Utah
  - Alexandria, Virginia
  - Virginia Beach, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- Tampere, Finland
- Galway, Ireland
- Oslo, Norway
- Sheffield, United Kingdom

REFERENCES:
- [Derived] Syage JA, Murray JA, Green PHR, Khosla C. Latiglutenase Improves Symptoms in Seropositive Celiac Disease Patients While on a Gluten-Free Diet. Dig Dis Sci. 2017 Sep;62(9):2428-2432. doi: 10.1007/s10620-017-4687-7. Epub 2017 Jul 28. PMID 28755266
- [Derived] Murray JA, Kelly CP, Green PHR, Marcantonio A, Wu TT, Maki M, Adelman DC; CeliAction Study Group of Investigators. No Difference Between Latiglutenase and Placebo in Reducing Villous Atrophy or Improving Symptoms in Patients With Symptomatic Celiac Disease. Gastroenterology. 2017 Mar;152(4):787-798.e2. doi: 10.1053/j.gastro.2016.11.004. Epub 2016 Nov 15. PMID 27864127